CLINICAL TRIAL: NCT01546688
Title: A Randomised, Double Blind, Placebo-controlled Study to Evaluate the Safety and Tolerability and to Explore the Efficacy of Zonisamide as add-on Therapy in Elderly Patients With Refractory Partial Seizures
Brief Title: A Study to Evaluate the Safety and Tolerability and Explore the Efficacy of Zonisamide as add-on Therapy in Elderly Patients With Refractory Partial Seizures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2090-E044-402; 2006-002516-10 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zonisamide at targeted daily doses of 100-500 mg/day (Active Comparator)
  Interventions: Drug: Zonisamide at targeted daily doses of 100-500 mg/day
- Placebo administered to match daily doses of 100-500 mg/day (Placebo Comparator)
  Interventions: Drug: Placebo administered to match targeted daily doses of 100-500 mg/day

INTERVENTIONS:
Drug: Zonisamide at targeted daily doses of 100-500 mg/day — Each group received 2 doses a day (in the morning and evening) during the Titration Period, once a day (in the evening) or BID during the Maintenance Phase, comprising 25 mg, 50 mg, or 100 mg of ZNS capsules
  Arms: Zonisamide at targeted daily doses of 100-500 mg/day
Drug: Placebo administered to match targeted daily doses of 100-500 mg/day — matching placebo
  Arms: Placebo administered to match daily doses of 100-500 mg/day

SUMMARY:
A two arm, randomized, double-blind study comparing zonisamide with placebo. The zonisamide arm will consist of 100 subjects and the placebo arm of 50 subjects. Study medication will be administered as an add-on treatment to the subject's current 1 or 2 anti-epileptic (AEDs).

ELIGIBILITY:
Key Inclusion Criteria:

1. Capable of maintaining a seizure daily diary or who have access to a caregiver who is prepared to complete this on the patient's behalf.
2. Able to complete the questionnaires used in this study.
3. Localization related epilepsy, with simple and/or complex partial seizures with or without secondary generalized seizures as defined by the International League Against Epilepsy (ILAE) criteria.
4. Have at least one well documented seizure in the 4 weeks preceding the Randomisation Visit (Visit 2) and are deemed to require additional AED medication.
5. Receiving at least one, but not more than two other marketed AEDs as concomitant medication, and the dosage should be stable for at least four weeks before the Screening Visit.

Key Exclusion Criteria:

1. Seizures attributed to metabolic causes (e.g., electrolyte disturbances, hyperglycaemia).
2. Seizures which could be attributed to use of a drug.
3. Presence of primary generalised epilepsies or seizures, such as absences, myoclonic epilepsies, Lennox-Gastaut syndrome.
4. A history of eating disorders or a body weight below 40 kg.
5. A history of blood dyscrasias.
6. A history of renal stones or having risk factors for nephrolithiasis such as a family history of nephrolithiasis or hypercalciuria.
7. An increased risk factor for rhabdomyolysis such as uncontrolled hypothyroidism, personal or family history of muscle disorders.
8. Taking concomitant medication associated with nephrolithiasis and medications increasing the risk of rhabdomyolysis.
9. Taking rifampicin or drugs with anticholinergic effects.
10. Taking carbonic anhydrase inhibitors or topiramate.
11. A history of pancreatitis.
12. A history of Stevens Johnson Syndrome.
13. Elevated levels of serum creatinine >165 Umol, or known severe hepatic impairment to the extent that the protocol dose titration schedule cannot be followed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Segieth, Study Director — Eisai Limited
Locations (36):
- Germany (7):
  - Klinik und Polyklinik fur Epileptologie, Bonn
  - Georg-August-Universiat Gottingen, Göttingen
  - Asklepiosklinik Barmbek, Hamburg
  - Clinical Research Hamburg, Hamburg
  - ZNS Hamburg, Hamburg
  - Universitaet Giessen / Marburg, Marburg
  - Neurologische, Siegen
- Hungary (8):
  - Semmelweis University - Neurology Dept., Budapest
  - Synexus Magyarorszag Kft., Budapest
  - National Institute of Neurosurgery, Budapest
  - County Hospital Kecskemet, Keskemet
  - B-A-Z County Hospital - Szuleszet-Nogyogyaszat, Miskolc
  - Sopron Medical SMO, Sopron
  - County Hospital of Tolna, Szeksz?rd
  - County Hospital of Zala, Zalaegerszeg
- Italy (7):
  - S.C. Neurologia - AO "G.Brotzu", Cagliari
  - Dip. Di neuroscienze - Centro Epilessie - Osp. Careggi, Florence
  - Dipartimento di Neuroscienze - Universita Federico II, Napoli
  - Centro Epilessia - Istituto Neurologico "Fondazione C. Mondino", Pavia
  - Centro per la Diagnosi e Cura dell'epilessia - Policlinico Universitario di Messina, Pavia
  - Dip.to Scienze Neurologiche - III Clinica Neurologica, Roma
  - Universita di Torino - Dipt. Neuroscienze, Torino
- Medisch Centrum Haaglanden - Lokatie Westeinde, VA Den Haag, Netherlands
- Poland (7):
  - Specjalistyczny Zaklad Opieki Zdrowotnej 'KONSYLIUM', Kalisz
  - Specjalistyczna Praktyka Lekarska, Katowice
  - NZOZ Centermed Gabinety ?lnolekarskie, Leszno
  - Przych. Specj. I chorob Zaw. Wsi Instytut Medyc. Wsi im. W. Chodzki, Lublin
  - Oddzia Neurologiczny, Wojewdzki Szpital Specjalistyczny, Olsztyn
  - NZOZ Centrum Medyczne HCP, Późna
  - Wielospecjalistyczna Lecznica 'Zycie', Warsaw
- Switzerland (3):
  - Clinical Investigation Unit; Inselspital, Bern
  - Spitalzentrum Biel, Biel
  - Epilepsie-Zentrum, Zurich
- United Kingdom (3):
  - Whipps Cross university Hospital, London
  - University Hospital of North Staffordshire, Stoke-on-Trent
  - The Royal Cornwall Hospital, Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects took matching doses of placebo during both the Titration Period and Maintenance Period.
- Zonisamide: Subjects started the Titration Period on a Total Daily Dose (TDD) of zonisamide 50mg (25mg capsules twice daily in the morning and evening) for a total of 8 weeks. Doses increased in 100mg increments up to a targeted TDD of 300mg with a range of 100mg to 500mg. Subjects entered the Maintenance Period on the same dose they were on at the end of the titration phase, taking the dose once daily (in the evening) or twice daily for a total of 8 weeks. Subjects were withdrawn if they required a TDD outside of the suggested range.
Period: Overall Study
Arm/Group | Placebo | Zonisamide
Started | 18 | 33
Completed | 15 | 28
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zonisamide | Total
Number analyzed (Participants) | 18 | 33 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population
  Years | 71.1 (4.61) | 72.5 (5.63) | 72.0 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population: All randomized subjects who received at least one dose of study medication.
  Participants
    Female | 11 | 19 | 30
    Male | 7 | 14 | 21
Race/Ethnicity, Customized [Number; unit: Participants] — Race. Safety Population.
  Participants
    White | 18 | 33 | 51
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity. Safety Population.
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 17 | 31 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in CVST of the FePsy Test (Mean Reaction Time) by Visit During Titration and Maintenance Period
Description: The Computer Visual Search Task (CVST) of the Ferrum Psyche (FePsy)measured cognition. A decrease from Baseline (negative change value) signifies an improvement in the mean reaction time of CVST.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Intent-to-Treat Population: All randomized subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | Zonisamide
Number analyzed (Participants) | 18 | 33
Seconds
  Week 4 | -3.448 (10.212) | -3.898 (13.149)
  Week 8 | -2.776 (9.984) | -0.650 (10.140)
  Week 12 | -7.223 (11.949) | -2.731 (14.084)
  Week 16 | -3.324 (14.995) | -5.102 (11.526)

2. Primary Outcome: Change From Baseline in Bond and Lader Visual Analogue Scale (VAS) Mood Sub-Scores for Sedation by Visit During Titration and Maintenance Period
Description: The Bond-Lader mood rating scale measured sedation, with scores ranging from 0 to 100. A high score reflects a high level of sedation.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Zonisamide
Number analyzed (Participants) | 18 | 33
Scores on a Scale
  Week 4 | -1.337 (22.2976) | 1.654 (16.4085)
  Week 8 | 7.688 (17.0998) | 1.990 (16.0172)
  Week 12 | 1.386 (13.6130) | -0.682 (18.0567)
  Week 16 | 2.502 (17.6228) | 3.943 (21.0086)

3. Secondary Outcome: Percent Change in Seizure Frequency From Baseline to the Last 28 Days of the Maintenance Period
Description: Seizure frequency was assessed by a seizure diary, maintained daily from Baseline, in which the subject recorded the occurrence of any seizure.
Time Frame: Baseline and Month 4
Population: Intent-to-Treat Population.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Zonisamide
Number analyzed (Participants) | 18 | 33
Percent Change | -100 [-100 to 433] | -100 [-100 to 50]

4. Secondary Outcome: Percentage of Responders During Last 28 Days of Maintenance Period
Description: Seizure frequency was assessed by a seizure diary, maintained daily from Baseline, in which the subject recorded the occurrence of any seizure. A responder is a subject who had at least a 50 percent or greater reduction in the seizure frequency of all seizures during the last 28 days of the Maintenance Period compared to the Baseline Period seizure frequency. Due to the exploratory nature of the objective for efficacy and the truncated study size, analysis of efficacy was based on observed cases, without imputation for missing data. As a result, there are some variations in sample sizes for efficacy at different visits, depending on if particular efficacy variables were missing for particular visits.
Time Frame: Baseline and Month 4
Population: Intent-to-Treat Population. Percentages are based on the number of subjects present in the Maintenance Phase.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Zonisamide
Number analyzed (Participants) | 15 | 28
Percentage of Participants
  Responders (Yes) | 62.5 | 75
  Non-Responders (No) | 12.5 | 14.3
  Missing | 25 | 10.7

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAE) were collected, and includes all Adverse Events (AE) with a start date on or after Day 1 and within 15 Days of last dose, including AEs with missing start dates. Participants were followed for up to 27 weeks.
Arm/Group | Placebo | Zonisamide
Serious Adverse Events (participants affected / at risk) | 1/18 | 6/33
Other Adverse Events (participants affected / at risk) | 8/18 | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Zonisamide (N=33)
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Vertebrobasilar insuffficiency (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Zonisamide (N=33)
Anxiety (Psychiatric disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Asparatate aminotransferase increased (Investigations) | 1 | 0
Asthenia (General disorders) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 4
Hypertension (Vascular disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Radicular syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No